CLINICAL TRIAL: NCT06776185
Title: Recurrence Patterns and Cost-Effectiveness of Robotic-assisted, Laparoscopic, and Open Liver Resection in BCLC 0/A Hepatocellular Carcinoma:
Brief Title: Recurrence Patterns and Cost-Effectiveness of Surgical Approaches in Early-Stage Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Chen Xiaoping (Other)
Responsible Party: Sponsor-Investigator, Chen Xiaoping, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: RLOCE-001
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: HCC - Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Robotic-assisted: RALR was conducted using a robotic platform, which allowed for precise dissection and 3D visualization. Robotic arms equipped with advanced energy devices facilitated delicate maneuvers, particularly in deep or difficult-to-access segments. A 3D liver model was displayed on the robotic console, enabling real-time reference during dissection. As with LLR, intraoperative ultrasound refined the tumor boundaries, and the Pringle maneuver was selectively applied when necessary.
  Interventions: Procedure: Liver Surgery
- Laparoscopic: LLR was performed using standard laparoscopic instruments, with the surgeon directly manipulating instruments for tumor resection. Intraoperative ultrasound was routinely used to confirm tumor boundaries and refine resection margins, particularly for tumors adjacent to major vascular structures. During parenchymal transection, energy devices such as laparoscopic bipolar coagulators or ultrasonic scalpels were used to minimize blood loss. The Pringle maneuver was available as needed to control bleeding.
  Interventions: Procedure: Liver Surgery
- Open Liver Resection: Open liver resection was typically performed through a right subcostal incision, extended to the midline if necessary to enhance liver access. The liver was mobilized by dividing surrounding ligaments, including the falciform, coronary, and triangular ligaments, to ensure optimal exposure of the tumor. Intraoperative ultrasound was used to confirm the exact tumor location, delineate resection margins, and detect any additional satellite nodules or vascular invasion not identified preoperatively. The Pringle maneuver, involving intermittent clamping of the portal triad, was selectively applied to control blood loss during parenchymal transection. Based on tumor characteristics, anatomical resections aimed to remove full segments, while non-anatomical resections focused on achieving negative margins (R0 resection) with minimal liver removal. Large tumors, central lesions, or cases requiring complex vascular reconstruction were typically managed with the open approach due to its direct a
  Interventions: Procedure: Liver Surgery

INTERVENTIONS:
Procedure: Liver Surgery — Minimally Invasive Liver Resection In both LLR and RALR, standardized preoperative planning with 3D imaging was utilized to assess tumor location, size, and proximity to vascular structures, enabling precise port placement. Typically, four to five trocar ports were inserted based on the tumor's location, with adjustments as needed

SUMMARY:
This study aims to investigate the recurrence patterns and cost-effectiveness of robotic-assisted, laparoscopic, and open liver resections in patients with early-stage (BCLC 0/A) hepatocellular carcinoma. By analyzing data from 3000 patients across 27 centers, the research evaluates recurrence-free survival, overall survival, and long-term economic impacts using metrics such as quality-adjusted life years (QALYs) and incremental cost-effectiveness ratios (ICERs). Findings will provide insights into optimal surgical approaches to improve patient outcomes and healthcare resource utilization.

ELIGIBILITY:
Inclusion Criteria:

* (1) HCC diagnosis confirmed by two independent radiologists using contrast-enhanced computed tomography (CT) and/or magnetic resonance imaging (MRI) combined with postoperative pathology; (2) BCLC stage 0 or A; and (3) curative liver resection

Exclusion Criteria:

* (1) concurrent malignancies in other organs; (2) diagnosis of combined hepatocellular-cholangiocarcinoma; (3) prior neoadjuvant or adjuvant treatment before liver resection; (4) recurrent HCC; (5) ruptured HCC; and (6) incomplete follow-up or missing data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This multicenter study included BCLC stage 0/A HCC patients who underwent RALR, LLR, or OLR across 27 centers from July 2017 to July 2019
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Recurrence-free Surival | 2017-01-01--2024-01-01

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No